CLINICAL TRIAL: NCT00544089
Title: Chromosomal and Morphological Structure of Mature and Immature Male Germ Cells and Recognition of IL-18 in Testicular Tissue of Azoospermic Men
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 37/06
Record Dates: First submitted 2007-10-14; First posted 2007-10-16 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2006-03

CONDITIONS: Infertility
Keywords: azoospermia FISH IL-18 TESTICULAR BIOPSY
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To develop a biotechnological assay which will be able to recognize germ cells of the spermatogenic lineand and to identify the chromosomal and morphological structure of mature and immature male germ cells, in cases of of sperm production disorders(azoospermic patients).

To recognize IL-18 in testicular tissue of azoospermic men compared to control group as it has been suggested that this cytokine may serve as a paracrine defense factor in the male gonad associated to spermatogenesis.

DETAILED DESCRIPTION:
A new biotechnological assay was developed by adapting an existing computerized system which scans cell morphology and chromosomal ploidy in the same cell of hematologic line using digital technology, to recognize germ cells of the testis by their morphology and cytogenetics. Testicular tissues which obtained from 15 men were enzymatically digested and the cells received were fixed on slides. The cells were stained by Giemsa May Grinwald staining and scanned automatically in a bright field for cell morphology. Fluorescence in situ hybridization (FISH) using centromeric probes for chromosomes X, Y and 18 was performed on the same slide after destaining. The cells were automatically scanned and classified according to the ploidy of the chromosome signals. The presence of IL-18 in the same men's testis was examined parallelly, by immunohistochimical staining using specific antibody for human IL-18.

ELIGIBILITY:
Inclusion Criteria:

* Non-obstructive azoospermic patients

Exclusion Criteria:

* Obstructive azoospermia

Ages: 22 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25907 (Actual)
Dates: Start 2006-03; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Ron-el, professor, Principal Investigator — Assaf-Harofeh Medical Canter
Locations (1):
- Infertility unit, Asaf-Harofeh Medical Center, Zrifin, Israel